CLINICAL TRIAL: NCT00073879
Title: Allogeneic Adoptive Immunochemotherapy For Treatment Of Renal Cell Carcinoma
Brief Title: Fludarabine, Cyclophosphamide, and Alemtuzumab in Treating Patients With Recurrent or Metastatic Renal Cell Carcinoma (Kidney Cancer) Undergoing Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Purpose: Treatment
Other Study IDs: CDR0000328247; BCM-H-8447
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Alemtuzumab; Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: alemtuzumab
Biological: graft-versus-tumor induction therapy
Drug: cyclophosphamide
Drug: fludarabine phosphate
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy. Sometimes the transplanted cells can reject the body's normal tissues. Alemtuzumab and tacrolimus may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of combining fludarabine and cyclophosphamide with alemtuzumab in treating patients who are undergoing allogeneic stem cell transplantation for recurrent or metastatic renal cell carcinoma (kidney cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of fludarabine, cyclophosphamide, and alemtuzumab in patients with recurrent or metastatic renal cell carcinoma undergoing HLA-matched allogeneic stem cell transplantation.

OUTLINE: This is a pilot, multicenter study.

* Conditioning: Patients receive fludarabine IV over 30 minutes on days -6 to -2, cyclophosphamide IV over 2 hours on days -6 and -5, and alemtuzumab IV on days -4 to -2.
* Allogeneic transplantation: Allogeneic stem cells are infused on day 0. Patients receive graft-vs-host disease prophylaxis with tacrolimus IV or orally for approximately 30 days.

Patients are followed weekly for 100 days and then at 6, 12, 18, 24, 36, 48, and 60 months after transplantation.

PROJECTED ACCRUAL: A total of 20 patients (10 with HLA-identical related donors and 10 with matched unrelated donors) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent or metastatic renal cell carcinoma
* Failed interleukin-2 (IL-2)-based therapy OR intolerant to IL-2
* Clinically evident and followable disease
* Availability of 1 of the following compatible donors:

  * Related HLA-identical or 1-Ag mismatched donor
  * Unrelated HLA-A, B, DRB1-matched donor

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Karnofsky 70-100%

Life expectancy

* No concurrent illness that severely limits life expectancy

Hematopoietic

* Not specified

Hepatic

* No episode of hepatitis within the past month
* No evidence of chronic active hepatitis or cirrhosis

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* LVEF at least 40%
* No uncontrolled arrhythmias
* No symptomatic cardiac disease

Pulmonary

* FEV_1, FVC, and DLCO at least 50% of predicted (unless due to metastatic disease)

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment related mortality | 100

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States